CLINICAL TRIAL: NCT02584114
Title: Brain Effects of Memory Training in Early Psychosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Lisa Buchy, Postdoctoral Fellow, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB15_2463
Record Dates: First submitted 2015-10-15; First posted 2015-10-22 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory training group (Experimental): The intervention is self-administration of 4 hours of memory training over 4 days per week, for 3 weeks (12 hours total). Memory training will be done with the Peak app for memory training http://www.peak.net.
  Interventions: Behavioral: Peak app for memory training
- Non-memory training group (Active Comparator): The intervention is self-administration of 4 hours of training of games that do not involve memory such as language and card games over 4 days per week, for 3 weeks (12 hours total).
  Interventions: Behavioral: Non-memory training group

INTERVENTIONS:
Behavioral: Peak app for memory training
  Arms: Memory training group
Behavioral: Non-memory training group
  Arms: Non-memory training group

SUMMARY:
Background: People with psychosis show profound deficits in memory. A new cognitive remediation therapy using an app on a computer or mobile phone to improve memory has been effective in this population, but the neurobiological effects are unknown.

Objectives: 1) To use functional magnetic resonance imaging (fMRI) to examine brain changes during a working memory task before and after a 12 hour memory training intervention on a computer or mobile phone, 2) To use diffusion tensor imaging (DTI) to examine white matter connecting prefrontal and parietal lobe before and after training.

Methods: 46 people with psychosis will be randomized to a computerized training of either memory training or a control condition of non-memory games (language/card games) and will self-administer 4 hours of training over 4 days per week, for 3 weeks (12 hours total). Memory training will be done with the Peak app http://www.peak.net. Imaging data will be gathered with a 3 Tesla scanner pre and post training.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and between the ages of 18 and 40
2. Able to understand and sign an informed consent document in English.
3. Meet diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or psychosis not otherwise specified.

Exclusion Criteria:

1. Impaired intellectual functioning (full-scale IQ<70).
2. Past or current history of a clinically significant central nervous system disorder that may contribute to psychotic symptoms or confound their assessment.
3. Current severe substance use disorder.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in functional Magnetic Resonance Imaging blood oxygen-dependent signal during working memory task performance before and after a 12 hour memory training intervention in people with early psychosis | 5 weeks
Change in diffusion tensor imaging measured change in fractional anisotropy during working memory task performance before and after a 12 hour memory training intervention in people with early psychosis | 5 weeks